CLINICAL TRIAL: NCT03029962
Title: Girl2Girl: Harnessing Text Messaging to Reduce Teenage Pregnancy Among LGB Girls
Acronym: Girl2Girl
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency); University of British Columbia (Other); City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1 TP2AH000035-01-00
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Teenage Pregnancy
Keywords: Teenage Pregnancy Prevention; LGB Girls; Text-Messaging; Information-Motivation-Behavioral Skills(IMB)Model

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental: Girl2Girl (Experimental): Girl2Girl is a 7-week teenage pregnancy prevention program delivered daily via text messaging to 14-18 year old females who self-identify as lesbian, bisexual, gay, or other sexual minority. In addition to program content, participants are paired with another participant (i.e., a Text Buddy) with whom they can text throughout the program to provide support; and an on-demand advice line, Girl2Genie, which shares information about sex, relationships, and the lesbian, gay, bisexual, transgender (LGBT) community.
  Interventions: Behavioral: Girl2Girl
- No Intervention: Health Lifestyle (No Intervention): The attention-matched control arm message content consists of information publicly available online related to living a healthy lifestyle. Content discussed includes: nutrition and sleep hygiene, self-esteem and body image, bullying, and drugs and alcohol. The control arm is 7-weeks in length (Week 7 is a review booster) and is delivered via text messaging. Messages are didactic and not tailored to user sexual experience. Additionally, the Text Buddy and G2Genie intervention program components are not available.

INTERVENTIONS:
Behavioral: Girl2Girl — Girl2Girl is a text messaging-based teenage pregnancy prevention program specifically for 14-18 year old LGB adolescent females. Content is guided by the Information-Motivation-Behavioral Skills (IMB) model and focuses on: HIV information, motivations to engage in HIV preventive behavior, communication skills, behavioral skills (e.g., using a condom; HIV testing); and healthy/unhealthy relationships. Behavioral skills content is reinforced using brief online videos. The intervention is 7 weeks long. A "booster" is delivered 12-weeks post-intervention end and reviews the topics covered in the intervention. Girl2Girl content is tailored based upon sexual experience (i.e., whether one is abstinent or sexually active) and whether one is same-sex or dually attracted.
  Arms: Experimental: Girl2Girl

SUMMARY:
The purpose of this study is to finalize and rigorously evaluate Girl2Girl, a novel text messaging-based teenage pregnancy prevention (TPP) program designed specifically for LGB women ages 14-18 years, nation-wide. The guiding theoretical model is the Information-Motivation-Behavioral Skills (IMB) Model, which has been used extensively and is associated with increases in TPP behavior.

DETAILED DESCRIPTION:
An estimated one in four teen women will become pregnant by the time she is 20 years of age. That said, significant disparity in rates exist for lesbian, gay, bisexual and other sexual minority women (LGB) versus non-LGB teen women: Research suggests that lesbian and bisexual teen women are between two and four times more likely to report having been pregnant than teen women who identified as exclusively heterosexual. Despite this compelling evidence that lesbian and bisexual adolescent women are at risk for teen pregnancy, programs tailored to the unique needs of adolescent LGB women are nonexistent. Evidence-based teen pregnancy prevention (TPP) programs targeting LGB teen women are urgently needed.

The Girl2Girl intervention text messaging-based TPP program designed specifically for LGB women ages 14-18 years, nation-wide. The investigators will test the intervention in a randomized control trial (RCT) of 840 LGB teenage women randomly assigned to either the intervention (n = 420) or control (n = 420) arms. Our primary efficacy outcome measures, measured at 12-months post-intervention, will be: (a) abstinence from penile-vaginal sex; (b) condom use during penile-vaginal sex, (c) use of other birth control methods during penile-vaginal sex, and (d) pregnancy.

If effective, Girl2Girl has promise to be quickly and cost-effectively implemented to scale to help to curb the spread of teenage pregnancy among women who identify as LGB.

ELIGIBILITY:
Inclusion Criteria:

* endorse a non-heterosexual sexual identity (i.e., lesbian/gay, bisexual, queer, questioning, unsure);
* be cisgender (i.e., be assigned a female sex at birth and endorse a female gender identity);
* be aged 14-18;
* in high school or equivalent (including those who did not finish school/dropped out);
* be English speaking;
* be exclusive owners of a cell phone with an unlimited text messaging plan;
* have used text messaging for at least six months;
* intend to have the same cell number for the next six months; and,
* be able to provide informed assent, including an acceptable score for "capacity to consent" and the self-safety assessment.

Exclusion Criteria:

* not having the capacity to assent
* not passing the self-safety assessment
* previously participating in another study activity (with the exception of the baseline and intervention end survey pilot tests)
* knowing someone who is already enrolled in the program
* non-cisgender

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — cisgender / female gender identity
Enrollment: 948 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Number of protected penile-vaginal sex acts | Post-intervention (about 20 weeks after randomization)
  The relative difference of protected penile-vaginal sex acts in the intervention versus control group at 12-months post-intervention
Number of participants who used other birth control methods | Post-intervention (about 20 weeks after randomization)
  The relative difference of teens who used birth control methods other than condoms (e.g., the pill, the patch) in the intervention versus control group at 12-months post-intervention
Number of participants who abstained from penile-vaginal sex | Post-intervention (about 20 weeks after randomization)
  The relative difference of abstinence (not engaging in vaginal sex) in the intervention versus control group at 12-months post-intervention

SECONDARY OUTCOMES:
Number of penile-vaginal sex acts during which a condom was used | immediate post-intervention end, 3-, 6-, 9-months post-intervention
  The relative difference of protected penile-vaginal sex acts in the intervention versus control group at immediate post-intervention end, 3-, 6-, and 9-months post-intervention
Number of participants who used other birth control methods | immediate post-intervention end, 3-, 6-, 9-months post-intervention
  The relative difference of teens who used birth control methods other than condoms (e.g., the pill, the patch) during penile-vaginal sex acts in the intervention versus control group at immediate post-intervention end, 3-, 6-, and 9-months post-intervention
Number of participants who abstained from penile-vaginal sex | immediate post-intervention end, 3-, 6-, 9-months post-intervention
  The relative difference of abstinence (not engaging vaginal sex) in the intervention versus control group at immediate post-intervention end, 3-, 6-, and 9-months post-intervention
Pregnancy | Across the 12 months post-intervention
  The percent of teens who have been pregnant since the beginning of the RCT in the intervention versus control group

OTHER OUTCOMES:
Intentions to use condoms | immediate post-intervention end, 3-, 6-, 9-, and 12-months post-intervention
  The percent of teens who intend to use condoms if they have penile-vaginal sex in the next year in the intervention versus control group
Intentions to use birth control other than condoms | immediate post-intervention end, 3-, 6-, 9-, and 12-months post-intervention
  The percent of teens who intend to use birth control methods other than condoms in the next year for the intervention versus control group

CONTACTS AND LOCATIONS:
Overall Officials: Michele L Ybarra, PhD, Principal Investigator — Center for Innovative Public Health Research
Locations (1):
- Center for Innovative Public Health Research, San Clemente, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ybarra ML, Parrilla JS, Wolowic J, Rosario M, Goodenow C, Saewyc E. A National, Qualitative Study of Sexual Decision Making by Teenage Girls who are Lesbian, Gay, Bisexual, or who have Another Nonheterosexual Identity. J Pediatr. 2020 Feb;217:177-183. doi: 10.1016/j.jpeds.2019.10.038. Epub 2019 Dec 13. PMID 31843216
- [Background] Doull M, Wolowic J, Saewyc E, Rosario M, Prescott T, Ybarra ML. Why Girls Choose Not to Use Barriers to Prevent Sexually Transmitted Infection During Female-to-Female Sex. J Adolesc Health. 2018 Apr;62(4):411-416. doi: 10.1016/j.jadohealth.2017.10.005. Epub 2017 Dec 28. PMID 29290373
- [Derived] Ybarra ML, Saewyc E, Rosario M, Dunsiger S. Subgroup Analyses of Girl2Girl, a Text Messaging-Based Teen Pregnancy Prevention Program for Sexual Minority Girls: Results from a National RCT. Prev Sci. 2023 Dec;24(Suppl 2):292-299. doi: 10.1007/s11121-023-01493-6. Epub 2023 Feb 8. PMID 36753043

DOCUMENTS (1):
  • Informed Consent Form (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT03029962/ICF_000.pdf